CLINICAL TRIAL: NCT05293613
Title: Extracorporeal Shock Wave Lithotripsy for Treatment of Large Pediatric Renal Pelvic Stone Burden More Than 2 cm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Khalaf Elsayed, resident doctor at urolrogy department sohag university hospital, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh_Med_22_03_04
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Determine the Efficacy and Safety of SWL in Renal Stones Larger Than 2 cm in Pediatric Age Group
MeSH Terms: interventions — Lithotripsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cases (Experimental)
  Interventions: Device: extracorporeal shock wave lithotripsy

INTERVENTIONS:
Device: extracorporeal shock wave lithotripsy — shock wave transmited from the device through patient body towards the stone to disintegrate it

SUMMARY:
Extracorporeal shock wave lithotripsy (SWL) was first described for pediatric nephrolithiasis in 1986; SWL has been a mainstay of treatment for both renal and ureteral calculi in children . SWL is currently regarded as first-line therapy for most renal and upper ureteral calculi <2.0 cm according to the EAU/ESPU guidelines . Meanwhile, the American Urological Association (AUA) considers SWL to be a first-line option along with URS for renal or ureteral calculi <2.0 cm, and a first-line option along with PNL for renal calculi >2.0 cm . The shock waves are better transmitted and spontaneous clearance of fragmented stones in pediatric kidneys is higher than adults' kidneys; thus, SWL treatment seems likely to be more successful in the pediatric population compared to the adult population .Younger age is associated with better stone clearance in children treated with SWL, and this is related mostly to increased ureteral compliance (shorter, more elastic and distensible) and shorter skin-to-stone distance .

ELIGIBILITY:
Inclusion Criteria:

* Age: 1 year - 5 years old. ( as children younger than 5 years old has shorter skin to stone distance & the option of endoscopic treatment of stones has is not feasible in this age group) Stone size: more than 2 cm & less than 3.5 cm. Stone location: renal pelvis & other calyces.

Exclusion Criteria:

* Age: less than 1 year & more than 5 years old. Stone size: less than 2 cm & more than 3.5 cm. Raised serum creatinine , coagulopathy. Distal urinary tract obstruction. Pulmonary or cardiac disease Anatomical abnormalities (UPJO, horses shoe kidney, ...)

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
stone free rate | 2 months
  degree of stone disintegration & expulsion form pediatric patient after going through Extracorporeal shock wave lithotripsy for treatment of large pediatric renal pelvic stone burden more than 2 cm

SECONDARY OUTCOMES:
complications associated with pediatric SWL | 2 months
  Study complications associated with pediatric SWL with large stone burden > 2cm

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Sultan S, Aba Umer S, Ahmed B, Naqvi SAA, Rizvi SAH. Update on Surgical Management of Pediatric Urolithiasis. Front Pediatr. 2019 Jul 3;7:252. doi: 10.3389/fped.2019.00252. eCollection 2019. PMID 31334207
- [Background] Tasian GE, Copelovitch L. Evaluation and medical management of kidney stones in children. J Urol. 2014 Nov;192(5):1329-36. doi: 10.1016/j.juro.2014.04.108. Epub 2014 Jun 21. PMID 24960469
- [Background] Gajengi AK, Wagaskar VG, Tanwar HV, Mhaske S, Patwardhan SK. Metabolic Evaluation in Paediatric Urolithiasis: A 4-Year Open Prospective Study. J Clin Diagn Res. 2016 Feb;10(2):PC04-6. doi: 10.7860/JCDR/2016/17265.7251. Epub 2016 Feb 1. PMID 27042515